CLINICAL TRIAL: NCT06186908
Title: Assessment of Saliva Galectin-7, Galectin-10 and MMP-9 Levels In Individuals With Different Periodontal Diseases
Brief Title: Evaluation of Salivary Gal-7, Gal-10 and MMP-9 Levels of Individuals With Different Periodontal Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ceren Koksal, Research Assistant at Periodontology, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-TDU-DİŞF-0015
Record Dates: First submitted 2023-12-17; First posted 2024-01-02 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Periodontal Diseases
MeSH Terms: conditions — Periodontal Diseases

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) samples of saliva were obtained from 60 systemically healthy non-smoker individuals with periodontitis (P, n=20), gingivitis(G, n=20) and healthy periodontium (S, n=20)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy periodontium (Experimental): Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining
- Gingivitis (Experimental): Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining
- Periodontitis (Experimental): Full-mouth clinical periodontal measurements recorded and saliva obtained.
  Interventions: Diagnostic Test: Saliva obtaining

INTERVENTIONS:
Diagnostic Test: Saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
The aim of this study is; detection of Galectin-10, Galectin-7, MMP-9 levels in saliva samples of periodontally healthy, gingivitis and periodontitis patients and the possible correlation between these values and clinical parameters of periodontal diseases. Materials and methods: Samples of saliva were obtained from 60 systemically healthy non-smoker individuals with periodontitis (P, n=20), gingivitis(G, n=20) and healthy periodontium (S, n=20). Full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL), bleeding on probing (BOP), gingival index (GI) and plaque index (PI) were also recorded. Enzyme-linked immunosorbent assay (ELISA) was used to determine Galectin-10, Galectin-7 and MMP-9 levels in the biological samples.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (The determination of healthy volunteers will be based on the statements of the patients in the anamnesis. No additional examinations will be made.)
* At least twenty permanent teeth in the mouth
* Non-smoker
* No medication for continuous use
* Those who have not used antibiotics, anti-inflammatory and systemic corticosteroid drugs in the last 6 months.
* Not in pregnancy or lactation period.
* For the periodontitis group that has not received periodontal treatment in the last 6 months
* For the periodontitis group; According to the evaluation made in 6 regions of each tooth, individuals with 30% or more bleeding on probing area, at least 2 teeth not adjacent to each quarter jaw with a depth of 5 mm or more and 4 mm or more attachment loss, coronal 1/3 and more on radiography (horizontal and / or vertical) bone loss
* For the gingivitis group; According to the evaluation made in 6 regions of each tooth, individuals with 10% or more bleeding on probing area, having a probing depth of less than 4mm and no attachment loss
* For healthy group; According to the evaluation made in 6 regions of each tooth,individuals with less than 10% bleeding on probing area, having a probing depth less than 4mm and no loss of attachment were included in the study.

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months
* Smokers are not included in the study

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-03-24 (Estimated)

PRIMARY OUTCOMES:
The total amount of Gal-10 in saliva | 24 hours after taking the clinical measurements at the first visit
  The total amount of Galectin-10 in saliva
The total amount of Gal-7 in saliva | 24 hours after taking the clinical measurements at the first visit
  The total amount of Galectin-7 in saliva
The total amount of MMP-9 in saliva | 24 hours after taking the clinical measurements at the first visit
  The total amount of Matrix metalloproteinase 9 in saliva

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Sağlam, Study Director — Izmir Katip Çelebi University
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF